CLINICAL TRIAL: NCT05805735
Title: Anti-Wrinkle Efficacy Study
Brief Title: Anti-Wrinkle Efficacy Study of an Eye-Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23.0076-27
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Aging; Wrinkle

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison
Masking Description: Blinding of sponsor label (de-branded product)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Face care product (Eye cream) (Experimental): Comparison between assessment times. Assessments will be performed before, after 2, 4 and 8 weeks of product application.
  Interventions: Other: Face care product (Eye cream)

INTERVENTIONS:
Other: Face care product (Eye cream) — The test material(s) will be cosmetic products to be applied around the eye region on both sides of the face daily. The test product will be applied twice daily in the morning and in the evening by the subjects

SUMMARY:
The purpose of this study is to assess the anti-aging and reduction of dark circles efficacy of a cosmetic product after 8 weeks of application.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female and male (approx. 10% male)
* Between 40 and 65 years of age
* Visible wrinkles in the periorbital regions in accordance with the study site's score of at least grade 3
* Dark circles according to self-assessment (not guaranteed on darker skin types)
* Healthy skin in the test areas
* Uniform skin color and no erythema or dark pigmentation (except dark cycles are still visible) in the test area

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension (if not adjusted with medication), cardiovascular diseases
* Insulin-dependent diabetes mellitus
* Any topical medication at the test area within the last 7 days prior to the start of the study and/or throughout the entire course of the study
* Documented allergies to face care or cleansing products
* Active skin disease at the test area
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, etc. at the test area that could influence the investigation
* Past cosmetic surgery procedure in the test area (e.g. laser, facelift)
* Cosmetic surgery procedure in the test area, e.g. IPL (Intensed Pulsed Light), botox, chemical peel, dermabrasion within the last 2 years prior to the start of the study
* Epilepsy
* Obesity with a BMI > 40
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. antiallergics) and/or within the last 7 days prior to the start of the study
* Medical treatment for wrinkle reduction (e.g. peeling with vitamin A or fruit acids) on the face within the last 2 weeks prior to the start of the study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Anti-wrinkle efficacy will be assessed in the periorbital regions wrinkles using DermaTOP. Parameters measured: Rz and Ra, representing mainly the rough structure (Rz) or the finer skin structure (Ra). | 8-weeks

SECONDARY OUTCOMES:
Change from baseline in skin firmness by Cutometer [mm] after 2, 4 and 8 weeks | 8-weeks
Change from baseline in skin elasticity by Cutometer after 2, 4 and 8 weeks | 8-weeks
Change from baseline in skin hydration (assessed on skin capacitance by Corneometer [a.u.]) after 2, 4 and 8 weeks | 8-weeks
Change from baseline in skin barrier function (assessed on transepidermal waterloss by Tewameter [g/(m²h)]) after 2, 4, 8-weeks | 8-weeks
Dark circles color in difference by ColorFace image analysis Clinical assessment of dark circle reduction around the eye area by trained grader | 8-weeks
Clinical assessment of dark circle reduction by trained grader | 8-weeks
Subjective Evaluation of product traits assessed via questionnaire after 2, 4 and 8 weeks | 8-weeks
Assessment of eye area puffiness by photo ranking by 3 trained graders | 8-weeks
Photo documentation of skin by ColorFace | 8-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Röck, Dipl. Biol, Principal Investigator — SGS proderm GmbH
Locations (1):
- proderm GmbH, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No